CLINICAL TRIAL: NCT01148810
Title: A Multi-centre, Double-blind, Placebo Controlled, Proof of Concept Study to Evaluate the Efficacy and Tolerability of BAF312 in Patients With Polymyositis and Dermatomyositis
Brief Title: Efficacy and Tolerability of BAF312 in Patients With Polymyositis and Dermatomyositis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was prematurely terminated due to enrollment challenges.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBAF312A2202; 2008-006311-21 (EudraCT Number)
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Polymyositis; Dermatomyositis
Keywords: Inflammatory muscle disease, Muscle weakness, Myositis, inflammatory myopathy, inclusion body myositis, skin rash, autoimmune, difficulty swallowing, dysphagia
MeSH Terms: conditions — Polymyositis; Dermatomyositis; Myositis; Muscle Weakness; Myositis, Inclusion Body; Exanthema; Deglutition Disorders | interventions — siponimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BAF312 (Experimental)
  Interventions: Drug: BAF312

INTERVENTIONS:
Drug: BAF312
  Arms: BAF312
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study determined the efficacy, safety, tolerability and the PK profile of BAF312, a novel immunomodulator, in polymyositis and dermatomyositis patients who were not responsive to traditional immunosuppressive and/or corticosteroid therapy. The study consisted of a 12 week, randomized, placebo controlled period, followed by another 12 weeks where all subjects received BAF312 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with disease at least 3 months before study
* Muscle weakness
* Received corticosteroids with or with out disease modifying antirheumatic drugs at least 3 months before study however not responding to this therapy

Exclusion Criteria:

* Other idiopathic inflammatory myopathies
* Myopathy other than polymyositis and dermatomyositis
* Patients with late stages of disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-06-15 (Actual); Primary Completion 2012-06-13 (Actual); Study Completion 2012-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Novartis Investigative Site, Boston, Massachusetts, United States
- Novartis Investigative Site, Prague, Czechia
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Novartis Investigative Site, Stockholm, Sweden
- Novartis Investigative Site, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was terminated after 18 patients had been enrolled, of which 14 were eligible for the primary efficacy analysis.
Groups:
- BAF312/BAF312: 2 tablets each of BAF312 5mg for oral administration in period 1 and 2 tablets each of BAF312 5mg in period 2
- Placebo/BAF312: 2 tablets of Placebo for oral administration in period 1 and 2 tablets each of BAF312 5mg in period 2
Period: Overall Study
Arm/Group | BAF312/BAF312 | Placebo/BAF312
Started | 8 | 10
Completed | 7 | 5
Not Completed | 1 | 5
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized set: all patients with Polymyositi/Dermatomyositis were enrolled and randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | BAF312/BAF312 | Placebo/BAF312 | Total
Number analyzed (Participants) | 8 | 10 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Randomized set
  Years | 51.4 (6.48) | 48.1 (15.57) | 49.6 (12.18)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Randomized set
  Participants
    Female | 4 | 7 | 11
    Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Responded to BAF312
Description: Preliminary clinical efficacy of BAF312 in patients with Polymyositis and dermatomyositis (PM/DM) using the International Myositis Assessment and Clinical Studies Group (IMACS) core set measures (including manual muscle testing, Physician's Global Activity Assessment (on a horizontal 10 cm visual analogue scale), Patient Global Activity Assessment (on a horizontal 10 cm visual analogue scale), Physical Function (Health Assessment Questionnaire), Muscle-associated Enzymes (CK, LDH, AST, ALT, aldolase) and Extra-Muscular Activity Assessment (Extra-muscular portion of Myositis Disease Activity Assessment Tool).
Time Frame: 12 weeks
Population: All patients with evaluable (or complete) PD measurement and no major protocol deviations which impact on PD data were included in the PD analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | BAF312/BAF312 | Placebo/BAF312
Number analyzed (Participants) | 8 | 8
Participants | 4 | 1
Statistical Analysis 1: Comparison: BAF312/BAF312 vs Placebo/BAF312; Test type: Superiority or Other; Bayesian analysis = 0.960; Probability that the difference (BAF312-Placebo) is greater than the threshold

2. Secondary Outcome: Number of Participants With a Change in Steroids Use After BAF312 Administration -Period 2
Time Frame: 12 weeks
Population: The Safety set included all patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | BAF312/BAF312 | Placebo/BAF312
Number analyzed (Participants) | 7 | 8
Participants
  Steroid reduction | 3 | 2
  Steroid increase1 | 1 | 2
  Steroid stable | 3 | 4

3. Secondary Outcome: Mean Plasma Concentrations of BAF312
Time Frame: baseline to end of trial (day 196)
Population: PK Analysis set in all disease types
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- BAF312: 2 tablets each of BAF312 5mg for oral administration in period 1 and 2 tablets each of BAF312 5mg in period 2
Arm/Group | BAF312
Number analyzed (Participants) | 15
ng/ml
  baseline: number analyzed (Participants) | 7
  baseline | 0 (0)
  Day 8: number analyzed (Participants) | 7
  Day 8 | 29.6 (25.7)
  Day 28 | 121 (73.1)
  Day 56 | 160 (62.3)
  Day 84 | 163 (77.3)
  Day 92: number analyzed (Participants) | 14
  Day 92 | 80.0 (83.3)
  Day 112: number analyzed (Participants) | 12
  Day 112 | 120 (49.0)
  Day 140: number analyzed (Participants) | 12
  Day 140 | 129 (65.5)
  Day 168: number analyzed (Participants) | 12
  Day 168 | 125 (61.9)
  Day 196 | 27.9 (79.2)

4. Secondary Outcome: Summary of CRP Levels
Description: Biomarkers reflecting efficacy in reducing systemic inflammatory components of the disease using serum markers such as C-reactive protein (CRP)
Time Frame: 12 weeks
Population: The Safety set included all patients who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | BAF312/BAF312 | Placebo/BAF312
Number analyzed (Participants) | 7 | 8
mg/L | 4.14 (3.870) | 6.38 (8.999)

5. Secondary Outcome: Efficacy in Modifying Health-related Quality of Life Measured by SF-36
Description: Short Form (36) Health Survey. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BAF312/BAF312 | Placebo/BAF312
Number analyzed (Participants) | 4 | 4
score on a scale
  Physical component score | 36.469 (7.5520) | 30.406 (14.5402)
  Mental component score | 44.449 (7.2194) | 49.063 (12.9628)

6. Secondary Outcome: Myositis Disease (MD) Activity Scores
Description: Myositis Disease Activity Scores. This is a combined tool that captures the physician's assessment of disease activity of various organ systems via the MYOSITIS INTENTION TO TREAT ACTIVITY INDEX (MITAX) and via the MYOSITIS DISEASE ACTIVITY ASSESSMENT VISUAL ANALOGUE SCALES (MYOACT) It rates the physician's overall assessment of the ongoing current disease activity for various systems by drawing a vertical mark on the 10-cm line for each system according to the following scale: left end of line = no evidence of disease activity, midpoint of line = moderate disease activity, and right end of line = extreme or maximum disease activity.
Time Frame: Week 12
Population: PD set in all disease types
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | BAF312/BAF312 | Placebo/BAF312
Number analyzed (Participants) | 8 | 10
cm
  Extramuscular global assessment: number analyzed (Participants) | 7 | 7
  Extramuscular global assessment | 1.51 (1.171) | 2.27 (1.607)
  Cutaneous disease activity: number analyzed (Participants) | 7 | 7
  Cutaneous disease activity | 1.11 (0.997) | 1.31 (1.999)

7. Secondary Outcome: Physician Global Activity Assessment
Description: Physician's overall assessment on a single 0-10 cm scale, where the higher score indicates higher disease activity.
Time Frame: Baseline, Week 12
Population: PD set in all disease types
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | BAF312/BAF312 | Placebo/BAF312
Number analyzed (Participants) | 8 | 10
cm
  Baseline: number analyzed (Participants) | 7 | 7
  Baseline | 4.88 (0.947) | 3.93 (1.557)
  Week 12: number analyzed (Participants) | 7 | 7
  Week 12 | 3.04 (1.816) | 4.91 (2.601)

8. Secondary Outcome: Patient Global Activity Assessment
Description: Patient's overall assessment on a single 0-10 cm scale, where the higher score indicates higher disease activity.
Time Frame: Baseline, Week 12
Population: PD set in all disease types
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | BAF312/BAF312 | Placebo/BAF312
Number analyzed (Participants) | 8 | 10
cm
  Baseline: number analyzed (Participants) | 8 | 8
  Baseline | 4.36 (1.986) | 4.75 (2.435)
  Week 12: number analyzed (Participants) | 7 | 7
  Week 12 | 4.50 (1.557) | 5.44 (2.421)

9. Secondary Outcome: Manual Muscle Testing (MMT) - 8 Score
Description: Manual Muscle Testing - 8 (MMT-8): Assessment of designated muscles manually by scoring each muscle from 0 to 10 where 0 is no strength and 10 is maximum strength. MMT- 8 includes 7 bilateral muscles (potential score 0-70 x 2) and one unilateral (axial) muscle (0-10 x1) so the total score ranges from 0 to 150 (maximum) where higher score indicates more strength.
Time Frame: Baseline, Week 12
Population: PD set in all disease types
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BAF312/BAF312 | Placebo/BAF312
Number analyzed (Participants) | 8 | 10
scores on a scale
  Baseline: number analyzed (Participants) | 8 | 8
  Baseline | 106.8 (12.56) | 106.6 (19.70)
  Week 12: number analyzed (Participants) | 7 | 7
  Week 12 | 115.0 (10.31) | 100.7 (23.75)

10. Secondary Outcome: Health Assessment Questionnaire
Description: Health Assessment Questionnaire (HAQ): This questionnaire is a patient reported outcome (PRO) which is self-administered by the patient. It is used to assess disability and comprises various categories related to usual daily activities. The patients report the amount of difficulty they have in performing some of these activities. Each question asks on a scale ranging from 0 to 3 if the categories can be performed without any difficulty (scale 0) up to cannot be done at all (scale 3). The total score is derived from these sub-scores and ranges from 0 to 3 where higher HAQ indicates more disability.
Time Frame: Baseline, Week 12
Population: PD set in all disease types
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | BAF312/BAF312 | Placebo/BAF312
Number analyzed (Participants) | 8 | 10
Score on a scale
  Baseline: number analyzed (Participants) | 8 | 8
  Baseline | 1.2969 (0.53426) | 1.2031 (0.90863)
  Week 12: number analyzed (Participants) | 7 | 7
  Week 12 | 1.2143 (0.41278) | 1.3929 (0.86129)

11. Secondary Outcome: Serum Levels of Muscle Enzymes
Time Frame: Baseline, Week 12
Population: PD set in all disease types
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | BAF312/BAF312 | Placebo/BAF312
Number analyzed (Participants) | 8 | 10
U/L
  Creatine Kinase - Baseline: number analyzed (Participants) | 8 | 8
  Creatine Kinase - Baseline | 204.0 (237.37) | 872.5 (1256.60)
  Creatine Kinase - Week 12: number analyzed (Participants) | 7 | 7
  Creatine Kinase - Week 12 | 153.7 (128.62) | 858.1 (1499.12)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 2 years.
Description: This was a randomized, double-blind, placebo-controlled trial followed by an open label extension period where all patients received BAF312.
Arm/Group | BAF312/BAF312 | Placebo/BAF312
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/16 | 3/10
Other Adverse Events (participants affected / at risk) | 12/16 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BAF312/BAF312 (N=16) | Placebo/BAF312 (N=10)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BAF312/BAF312 (N=16) | Placebo/BAF312 (N=10)
Palpitations (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Macular oedema (Eye disorders) | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Bronchitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Tinea versicolour (Infections and infestations) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 2
Sciatica (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Mechanical urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
The study was terminated due to new clinical data from overall BAF312 program (<10 mg/day already have optimal pharmacodynamic effect & clinical efficacy). There was no safety concern testing 10 mg BAF312 that would have required study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.